CLINICAL TRIAL: NCT05152524
Title: Distal Ischemic Stroke Treatment With Adjustable Low-profile Stentriever
Acronym: DISTALS
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rapid Medical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CLN-TR13-001
Record Dates: First submitted 2021-09-26; First posted 2021-12-10 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Ischemic Stroke; Neovascularization
MeSH Terms: conditions — Ischemic Stroke; Neovascularization, Pathologic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Treatment (Experimental): Mechanical thrombectomy with Tigertriever 13 EVT + MM (without thrombolysis).
  Interventions: Device: Tigertriever 13
- Control (No Intervention): Medical Management alone (without thrombolysis).

INTERVENTIONS:
Device: Tigertriever 13 — patients presenting within 24 hours of onset with an ischemic stroke with disabling neurological deficits due to a primary distal vessel occlusion (DVO) will be treated with the Tigertriever 13 device.
  Arms: Treatment

SUMMARY:
The objective of the DISTALS Study is to evaluate the safety and effectiveness of the Tigertriever 13 Revascularization Device in restoring blood flow in the neurovasculature by removing thrombus in patients presenting within 24 hours of onset with an ischemic stroke with disabling neurological deficits due to a primary distal vessel occlusion (DVO), as compared to medical management.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-85 years old.
2. Pre-stroke mRS ≤2.
3. Disabling presenting deficits that localize to the territory of the distal vessel occlusion. Disabling deficits are deficits that, if unchanged, would prevent the subject from performing basic activities of daily living (i.e., bathing, ambulating, toileting, hygiene, and eating) or returning to work.
4. NIHSS 4-24, or NIHSS 2-24 for patients with aphasia and/or hemianopia.
5. Perfusion lesion (Tmax >4.0 seconds) volume ≥10 cc on CTP or MR PWI within the territory of the anterior cerebral artery (ACA) segments, a non-dominant or co-dominant M2 middle cerebral artery (MCA) segment, an M3 MCA, or the posterior cerebral artery (PCA) segments.
6. Occluded distal vessel diameter ≥1.5 mm as measured on CTA or MRA.
7. Ischemic core lesion (rCBF<30% on CTP or ADC <620 on MR DWI) in ≤50% of the perfusion lesion volume.
8. Study treatment can be initiated within 24 hours of last known well time (last known time without current stroke symptoms).
9. Signed informed consent by patient or legally authorized representative.
10. Subject is not eligible for intravenous thrombolysis within 3 hours from stroke onset per FDA label and American Heart Association/American Stroke Association national guidelines. (Note: administration of intravenous thrombolytics should not be avoided or delayed in order to achieve participation in this study.)

Exclusion Criteria:

1. Evidence of acute brain hemorrhage on CT and/or MRI at admission.
2. Use of any other intra-arterial (IA) recanalization device prior to the Tigertriever 13 in the target vessel, including aspiration catheter.
3. The DVO is a secondary distal occlusion that occurred during a large vessel occlusion (LVO) thrombectomy procedure.
4. Excessive tortuosity or stenosis that is anticipated to prevent placement of the microcatheter in the target vessel. Tortuosity or stenosis will be determined on CTA or MRA prior to randomization.
5. Evidence of tandem occlusion in the cervical internal carotid artery (ICA), intracranial ICA, M1 MCA, dominant M2 MCA, vertebral artery (VA) or basilar artery (BA) on CTA or MRA.
6. Evidence of dissection in the extra or intracranial cerebral arteries.
7. Evidence of bilateral acute stroke or acute stroke in multiple territories (e.g., bilateral anterior circulation, anterior/posterior circulation).
8. Prior stroke in the last 3 months.
9. Anticipated inability to obtain 3-month follow-up assessments.
10. Females who are pregnant or breastfeeding.
11. Renal failure with serum creatinine >3.0 or Glomerular Filtration Rate (GFR) <30.
12. Pre-procedural severe sustained hypertension with SBP >220 and/or DBP >120.
13. Pre-procedural glucose <50 mg/dl (2.78 mmol/L) or >400 mg/dl (22.20 mmol/L).
14. Pre-procedural coagulation factor deficiency or oral anti-coagulant therapy with an international normalized ratio (INR) of more than 1.7.
15. Treatment with heparin within 48 hours with a partial thromboplastin time more than two times the laboratory normal.
16. Treatment with a direct oral anticoagulant (DOAC) within 48 hours.
17. Platelet count of less than 50,000/uL.
18. History of severe allergy to contrast medium, nickel, or Nitinol.
19. Known current use of cocaine at time of treatment.
20. Known or suspected cerebral vasculitis.
21. Known hemorrhagic diathesis.
22. Aneurysm in target vessel.
23. Intracranial tumor (apart from small meningioma, ≤2 cm in diameter).
24. Ongoing seizure due to stroke.
25. Evidence of active systemic infection.
26. Known cancer with metastases.
27. Suspicion of aortic dissection, septic embolus, or bacterial endocarditis.
28. Subject already participating in another study of an investigational treatment device or treatment.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 168 (Estimated)
Dates: Start 2022-03-25 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Successful reperfusion (CTP or MR PWI*) without sICH**. | 24±6 Hours post randomization
  *Successful reperfusion is defined as >50% reduction in substantial hypoperfusion (Tmax >4 seconds) volume between baseline and 24 ±6 hours of randomization.
  **sICH shall be defined as any parenchymal hematoma type 2, remote intracerebral hemorrhage, subarachnoid hemorrhage, or intraventricular hemorrhage that is the predominant cause of ≥4 point NIHSS deterioration at 24 ±6 hours of randomization.

SECONDARY OUTCOMES:
All cause mortality at 90 days. | 90 days post randomization.
  All cause mortality at 90 days.
Any asymptomatic intracranial hemorrhage within 24±6 hours of randomization. | 24±6 hours of randomization.
  Any asymptomatic intracranial hemorrhage within 24±6 hours of randomization.
Device/procedure related serious adverse events (SAEs). | 90 days post randomization.
  Device/procedure related serious adverse events (SAEs).
Unanticipated adverse device effect (UADEs). | During procedure
  Unanticipated adverse device effect (UADEs).
Volume of penumbral tissue salvaged at 24±6 hours of randomization (CTP or MR DWI/PWI). | 24±6 hours post randomization.
  Volume of penumbral tissue salvaged at 24 ±6 hours of randomization (CTP or MR DWI/PWI).
Successful reperfusion at 24 hours, defined as >50% reduction in substantial hypoperfusion (Tmax >4 seconds) volume between baseline and 24 ±6 hours of randomization (assessed in both Treatment and Control arms). | 24±6 hours post randomization
  Successful reperfusion at 24 hours, defined as >50% reduction in substantial hypoperfusion (Tmax >4 seconds) volume between baseline and 24 ±6 hours of randomization (assessed in both Treatment and Control arms).
Successful reperfusion (eTICI ≥2b50) rate in the distal occluded vessel after Tigertriever 13 mechanical thrombectomy (assessed in Treatment arm only). | 24±6 hours Post procedure
  Successful reperfusion (eTICI ≥2b50) rate in the distal occluded vessel after Tigertriever 13 mechanical thrombectomy (assessed in Treatment arm only).
modified Rankin Scale (mRS) score | 90 days post randomization
  Level of global disability at 90 days measured by the modified Rankin Scale (mRS) shift (tetrachotomized: 0, 1, 2, 3-6). Minimum score: 0; Maximum score: 6. Lower scores reflects a better clinical outcome, and higher scores reflects worse clinical outcome.
National Institutes of Health Stroke Scale (NIHSS) shift | 4 days post procedure
  NIHSS change from Baseline to Day 4. Minimum score: 0; Maximum score: 42. Lower scores reflects a better clinical outcome, and higher scores reflects worse clinical outcome.
EQ-5D score | 90 days post randomization
  Health-related quality of life at 90 days - EQ-5D. Minimum score: 1; Maximum score: 9. Lower scores reflects a better clinical outcome, and higher scores reflects worse clinical outcome.
MoCA: Montreal Cognitive Assessment | 90 days post randomization
  Cognitive function at 90 days. Minimum score: 0; Maximum score: 30. Higher scores reflects a better clinical outcome, and Lower scores reflects worse clinical outcome.

CONTACTS AND LOCATIONS:
Locations (20):
- United States (14):
  - Lakewood Regional Medical Center, Los Angeles, California
  - Los Robles, Thousand Oaks, California
  - WellStar Research Institute, Marietta, Georgia
  - Advocate Aurora Research Institute,, Chicago, Illinois
  - Corewell Health (Spectrum), Grand Rapids, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - University of Buffalo, Buffalo, New York
  - NYU Langone Health, New York, New York
  - Mount Sinai, New York, New York
  - Stony Brook University, Stony Brook, New York
  - Mercy Health, Toledo, Ohio
  - Semmes Murphey Foundation, Memphis, Tennessee
  - Valley Baptist Medical Center, Harlingen, Texas
  - Texas Stroke Institute, Plano, Texas
- CUB Hôpital Erasme, Brussels, Belgium
- Germany (4):
  - Universitätsklinikum Bonn, Bonn
  - Alfreid Krupp, Essen
  - Universitätsklinikum Schleswig-Holstein, Kiel
  - St. Lukas hospital, Radprax, Solingen
- Orebro University Hospital, Örebro, Sweden

IPD SHARING:
Plan to Share IPD: No